CLINICAL TRIAL: NCT06574698
Title: Adding Of Naxitamb In Induction Therapy For High Risk Neuroblastoma: A Prospective, Single-Arm Clinical Study
Brief Title: Adding Of Naxitamb In Induction Therapy For High Risk Neuroblastoma
Status: Recruiting | Type: Observational
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Principal Investigator, Tianyou Yang, Chief Surgeon of Pediatric surgical oncology, Guangzhou Women and Children's Medical Center
Other Study IDs: neuroblastoma 2024
Record Dates: First submitted 2024-08-18; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Neuroblastoma; GD2 Antibody (Naxitamab)
MeSH Terms: conditions — Neuroblastoma | interventions — naxitamab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- High risk Neuroblastoma: High risk Neuroblastoma
  Interventions: Drug: Addition of anti-GD2 immunotherapy (Naxitamab) at the stage of induction chemotherapy

INTERVENTIONS:
Drug: Addition of anti-GD2 immunotherapy (Naxitamab) at the stage of induction chemotherapy — Addition of anti-GD2 immunotherapy (Naxitamab) at the stage of induction chemotherapy

SUMMARY:
To explore the efficacy of adding anti-GD2 immunotherapy (Naxitamab) at the stage of induction chemotherapy for newly diagnosed high risk neuroblastoma patients. To investigate wether anding Naxitamab in the induction phase will improve the response rate at the end of induction therapy and further improve the overall survival rate.

ELIGIBILITY:
Inclusion Criteria:

Neuroblastoma patients who meet certain criteria are eligible for enrollment in the following stages of diagnosis:

1. Children with newly diagnosed stage 4 neuroblastoma according to the International Neuroblastoma Staging System (INSS) who meet the following criteria are eligible for enrollment: i. Age > 18 months (> 547 days) regardless of biological characteristics; or ii. Age 12-18 months (365-547 days), with one of the following three unfavorable biological characteristics (MYCN amplification, pathological type of poor histopathological prognosis, and/or DNA index = 1); or iii. MYCN amplification (MYCN signal increase > 4 times compared to reference signal) regardless of age or other biological characteristics.
2. Children with newly diagnosed stage 3 INSS neuroblastoma who meet the following criteria are eligible for enrollment: i. MYCN amplification (MYCN signal increase > 4 times compared to reference signal) regardless of age or other biological characteristics; or ii. Age > 18 months (> 547 days), with pathological type of poor histopathological prognosis regardless of MYCN status.
3. Children with newly diagnosed stage 2A/2B INSS neuroblastoma with MYCN amplification (MYCN signal increase > 4 times compared to reference signal) regardless of age or other biological characteristics. The subject must be aged ≤ 21 years at the time of initial diagnosis, and must be aged > 12 months at the time of enrollment.

Exclusion criteria:

Infants less than 1 year old, those aged 12-18 months, INSS stage 4, and all INSS stage 3 patients with favorable biological characteristics (i.e., non-amplified MYCN, good pathological histopathological prognosis, and DNA index >1) are not eligible.

Subjects who have received immunosuppressive treatment (excluding local steroids) within the last 4 weeks prior to enrollment. Subjects who are currently receiving any investigational drug.

Any other medical condition that, in the opinion of the investigator, may interfere with the interpretation of results or affect the subject's ability to provide informed consent, the legal guardian's ability to provide informed consent, and the subject's cooperation and participation in the study, including but not limited to malabsorption syndrome, mental illness, or substance abuse. Subjects with significant comorbidities (any serious medical condition unrelated to cancer or its treatment that is not covered by the detailed exclusion criteria and is expected to interfere with the investigation drug(s) action or significantly increase the severity of the trial treatment toxicity)

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Newly Diagnosed High risk Neuroblastoma
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
The number of the patients of VGPR or CR at the end of induction therapy | 5 years
  Measured by cross-sectional computed tomography (CT) or magnetic resonance imaging (MRI) imaging and/or by methyl iodobenzylguanidine (MIBG) or positron emission tomography (PET) scans and bone marrow (BM) responses, evaluated according to the 1993 International Neuroblastoma Response Criteria (INRC), and compared with relevant historical control groups.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 5 years
  According to the International Neuroblastoma Response Criteria (INRC) of 1993 and 2017, the proportion of complete or partial responses was calculated in newly diagnosed high-risk group patients with neuroblastoma who received standard induction therapy. The disease status was evaluated by CT or MRI and/or MIBG or PET scans and bone marrow aspiration. After two courses of treatment, the proportion of complete or partial responses was calculated in newly diagnosed high-risk group patients with neuroblastoma who received standard induction therapy after two courses of treatment were completed.
The number of days a patient survives | 3 years after the last patient was enrolled
  The overall survival (OS) of patients receiving standard-induced chemotherapy and GD2 antibody combination therapy.
The number of days the patient survive without relapse or progression | 3 years after the last patient was enrolled
  The event-free survival (EFS) of patients receiving standard-induced chemotherapy and GD2 antibody combination therapy.
The objective response rate (ORR) after 6 cycles of treatment. | 5 years
  The objective response rate (ORR) after 6 cycles of treatment.
The number of patients with adverse events related to treatment | 5 years
  The number of patients with adverse events related to treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Women And Children's Medical Center, Guanzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No